CLINICAL TRIAL: NCT00184522
Title: Aflurax Versus Nexium Given on Demand to Patients With Gastro-esophageal Reflux Disease.
Brief Title: On Demand Treatment of Reflux Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Ferrosan AS (Industry)
Responsible Party: Professor MD Per Farup, Norwegian University of science and technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SLV 02-01973
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2005-09

CONDITIONS: Gastroesophageal Reflux
Keywords: Gastroesophageal Reflux; Esomeprazole; Drug treatment
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — idoflux; Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aflurax (Experimental): pectin-containing natural product
  Interventions: Drug: Aflurax
- esomeprazole (Nexium) (Active Comparator): esomeprazole (Nexium)
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: Aflurax
  Other Names: Pectin-containing nature product
  Arms: Aflurax
Drug: esomeprazole
  Other Names: Nexium
  Arms: esomeprazole (Nexium)

SUMMARY:
A comparison of the effect of on demand treatment with a pectin-containing natural product (Aflurax) with that esomeprazole (Nexium)

DETAILED DESCRIPTION:
A randomized, controlled, open trial comparing the symptomatic effect of a pectin-containing product (Aflurax) with that of esomeprazole (Nexium 20 mg) given on-demand for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

Mild and moderate reflux symptoms Age > 17 years Informed consent -

Exclusion Criteria:

Other conditions that might explain the symptoms Abuse of drugs or alcohol

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2002-08; Primary Completion 2004-11 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Symptomatic relief

SECONDARY OUTCOMES:
Overall satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Per G Farup, PhD, Study Chair — Norwegian University of Science and Technology
Locations (9):
- Norway (9):
  - Gjøvik Specialist Centre, Gjøvik
  - Sykehuset Innlandet HF, Gjøvik, Gjøvik
  - Sykehuset Innlandet HF, Hamar, Hamar
  - Sykehuset Innlandet HF, Kongsvinger, Kongsvinger
  - Sykehuset Innlandet HF, Lillehammer, Lillehammer
  - Helse Nord-Møre og Romsdal, Molde
  - Mosjøen sykehus, Mosjøen
  - Helse Nord-Trøndelag, Namsos
  - Sykehuset Innlandet HF, Tynset, Tynset

REFERENCES:
- [Result] Farup PG, Heibert M, Hoeg V. Alternative vs. conventional treatment given on-demand for gastroesophageal reflux disease: a randomised controlled trial. BMC Complement Altern Med. 2009 Feb 24;9:3. doi: 10.1186/1472-6882-9-3. PMID 19236727